CLINICAL TRIAL: NCT04002050
Title: Cognitive Behaviour Therapy With Mindfulness Course for Building Workplace Resilience: A Pilot Randomized Controlled Trial
Brief Title: Creating Resilient Workplaces Study
Acronym: CReW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Jitender Sareen, Professor of Psychiatry, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019:165
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: PTSD; Anxiety Disorders; Depression; Stress Disorders, Posttraumatic
Keywords: Resilience; Workplace Engagement; Public Safety Personnel; Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Stress Disorders, Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBTm Course Intervention (Active Comparator): Participants placed in the intervention group will receive the CBTm Course. The CBTm Course consists of 5 classes, 90 minutes each, and held in-person on a weekly basis.
  Interventions: Behavioral: Cognitive Behavioural Therapy with Mindfulness Course
- Comparison Group (No Intervention): Participants in the comparison group will not receive the intervention during the study, but will be offered intervention once the study has been completed (i.e. 3 month waiting-period). However, in the event that a stressful situation arises while a participant is placed in the comparison group, the participant may seek assistance from the usual mental health supports offered through their respective occupational organizations, EAP programs, and other programs in the community. Following completion of the study, participants in the comparison group will be invited to attend the CBTm Course.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy with Mindfulness Course — The Cognitive Behaviour Therapy with Mindfulness (CBTm) Course for Public Safety Personnel is a brief psychoeducational course consisting of 5 classes (90 minutes each) occurring on a weekly basis. The CBTm course addresses the fundamentals of CBT and provides participants with practical strategies for managing stress (such as relaxation strategies, cognitive restructuring, goal setting, behavioural activation, and exposure therapy).
  Arms: CBTm Course Intervention

SUMMARY:
The proposed study aims to understand the impact of a 5-Class CBTm Course on variables contributing to workplace resilience among Public Safety Personnel (PSP). This involves examining the impact of the CBTm Course on prevention of PTSD and related conditions among PSPs. This research project will be undertaken using a randomized-controlled trial design. Questionnaires will be completed 1) before taking the course, 2) during the course, 3) after the course, and 4) at three-month follow-up.

DETAILED DESCRIPTION:
The current proposal plans to implement and evaluate a CBT intervention for building workplace resilience by preventing symptoms of PTSD and related conditions in Public Safety Personnel (i.e., police officers, firefighters, paramedics, emergency communications, and correctional officers), in Manitoba, Canada. The intervention used in this study is the Cognitive Behaviour Therapy with Mindfulness (CBTm) Course.

Participants will be randomized into either the intervention group (CBTm) arm or the comparison arm. Participants placed in the intervention arm will be invited to immediately participate in the CBT intervention. Participants in the comparison arm will be placed on a 3-month waiting-list and will be invited to attend the CBT intervention following completion of the study. While placed in the comparison arm, participants may access the usual mental health supports that are normally offered through their respective occupational organizations, EAP programs, and other programs in the community.

Those who do not meet eligibility criteria will not be enrolled into the study, but will still be invited to attend the CBTm classes as space allows. Ineligible participants will not be randomized and their data will not be used in our analysis of the trial.

The Cognitive Behaviour Therapy with Mindfulness (CBTm) Course for Public Safety Personnel is a brief psychoeducational course consisting of 5 classes (90 minutes each) occurring on a weekly basis. The CBTm course addresses the fundamentals of CBT and provides participants with practical strategies for managing stress (such as relaxation strategies, cognitive restructuring, goal setting, behavioural activation, and exposure therapy). The sessions will be facilitated by a mental health-professional (i.e. psychiatrist, psychologist, and/or social worker).

Participants will complete self-report evaluation forms at baseline, weekly at CBTm Classes 1 to 5, post-intervention at 6 weeks, and follow-up at 3 months. They will be asked to complete the following measures: (1) Modified DSM-5 Self-Rated Level 1 Cross-Cutting Measure - Adult, (2) Generalized Anxiety Disorder 7-item, (3) Patient Health Questionnaire 9-item (PHQ-9), (4) Session Evaluation questionnaire, (5) Homework Evaluation Form, (6) Post-Traumatic Stress Disorder Checklist for the DSM-5 (PCL-5) with Life Events Checklist (LEC-5) and Criterion A, (7) Connor-Davidson Resilience Scale 10 item (CD-RISC 10), (8) Client Satisfaction Questionnaire (CSQ-8), (9) Short Form-12 (SF-12), (10) Drop out Form, (11) Five Facet Mindfulness Questionnaire 15-Item (FFMQ-15), (12) Perceived Stress Scale, (13) Utrecht Work Engagement Scale 9-Item (UWES-9), and (14) Service Utilization Follow Up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Employed and on active duty as a police officer, firefighter, paramedic, dispatcher, or corrections officer
3. Employed in Manitoba

Exclusion Criteria:

1. Diagnosed by a psychologist or psychiatrist with a mental health disorder in the past 6 months
2. A history of mental health service use related to a mental disorder in the past 6 months
3. PCL-5 score ≥37
4. PHQ-9 score ≥10
5. GAD-7 score ≥10
6. Suicidal ideation in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Changes in PTSD Symptoms | To be completed at Baseline, at CBTm Classes at week 1,2,3,4,5, post-intervention at 6 weeks, and follow-up at 3 months.
  To examine the impact of the CBTm Course on symptoms of PTSD as measured by the Posttraumatic Stress Disorder Checklist for the DSM-5 (PCL-5). A 10% change in score on this measurement tool is considered clinically significant.
Changes in Anxiety Symptoms | To be completed at Baseline, at CBTm Classes at week 1,2,3,4,5, post-intervention at 6 weeks, and follow-up at 3 months.
  To examine the impact of the CBTm course on symptoms of anxiety as measured by the Generalized Anxiety Disorder 7 Item Scale (GAD-7). This questionnaire objectively determines initial symptom severity and monitors symptom changes/effect of treatment over time. Each item is scored on a scale of "0" (not at all) to "3" (nearly every day). Scores of 5, 10, and 15 are used as the cut-off points for mild, moderate and severe anxiety, respectively.
Changes in Depressive Symptoms | To be completed at Baseline, at CBTm Classes at week 1,2,3,4,5, post-intervention at 6 weeks, and follow-up at 3 months.
  To examine the impact of the CBTm course on symptoms of depression as measured by the Patient Health Questionnaire 9-item (PHQ-9). This questionnaire objectively determines initial symptom severity and monitors symptom changes/effect of treatment over time. Each item is scored on a scale of "0" (not at all) to "3" (nearly every day). Scores of 5, 10, and 15 are used as the cut-off points for mild, moderate and severe depression, respectively.
Changes in Resilience Level. | To be completed at Baseline, at CBTm Classes at week 1,2,3,4,5, post-intervention at 6 weeks, and follow-up at 3 months.
  To examine the impact of the CBTm Course on resilience as measured by the Connor-Davidson Resilience Scale 10 (CD-RISC10). This questionnaire is used to rate an individual's resilience on a scale of 1 - 40 with a higher score reflecting a higher level of self-identified resilience.

SECONDARY OUTCOMES:
Changes in Physiological and Mental Health Symptoms | To be completed at Baseline, CBTm Class in week 3, post-intervention at week 6, and follow-up at 3 months.
  To examine the impact of the CBTm Course on physiological and mental health symptoms as measured by the Short Form 12 (SF-12). The total score is compared to the mean scores of the general population to give ratings of above average, average and below average.
Changes in Perceived Stress Levels | To be completed at Baseline, CBTm Class in week 3, post-intervention at week 6, and follow-up at 3 months.
  To examine the impact of the CBTm Course on perceived levels of stress as measured by the Perceived Stress Scale. This scale classifies perceived stress levels into low (scores of 0-13), moderate (score of 14-26) and high stress (score of 27- 40).
Evaluation of Client Satisfaction | To be completed at the 5th CBTm Class at Week 5 of the intervention.
  To examine client satisfaction of the CBTm Course as measured by the Client Satisfaction Questionnaire. Higher total scores indicate greater satisfaction.
Changes in the ability to engage in Mindfulness | To be completed at Baseline, CBTm Class in week 3, post-intervention at week 6, and follow-up at 3 months.
  To examine the impact of the CBTm Course on one's ability to engage in mindfulness as measured by the 15-Item Five Facet Mindfulness Questionnaire. The five areas of mindfulness measured are: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Higher total/sub-scale scores indicate increased engagement in mindfulness.
Changes in Work Engagement | To be completed at Baseline, CBTm Class in week 3, post-intervention at week 6, and follow-up at 3 months.
  To examine the impact of the CBTm Course on work engagement as measured by the 9-Item Utrecht Work Engagement Scale. The measure is scored over three dimensions: vigor, dedication, and absorption. Higher total scores are negative correlates of burnout.
Service Utilization Follow Up | To be completed at the 3 month follow-up.
  To determine whether any participants received service or treatment for emotional, alcohol or drug problems while enrolled in the study, which are confounding variables that may potentially affect the study's results

CONTACTS AND LOCATIONS:
Overall Officials: Shay-Lee Bolton, PhD, Study Director — University of Manitoba; Dov Millstone, MPH, Study Director — University of Manitoba; Jitender Sareen, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba Department of Psychiatry, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No